CLINICAL TRIAL: NCT02449304
Title: Evaluation of Feasibility and Effectiveness of 4th Generation Bipolar Radiofrequency Endometrial Ablation Device: a Cohort Study
Brief Title: Evaluation of 4th Generation Bipolar Radiofrequency Endometrial Ablation Device
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Birmingham Women's NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Thomas Justin Clark, Professor, Birmingham Women's NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BirminghamWHC
Record Dates: First submitted 2015-05-13; First posted 2015-05-20 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Heavy Menstrual Bleeding
Keywords: endometrial ablation, heavy menstrual bleeding, novosure
MeSH Terms: conditions — Menorrhagia | interventions — Endometrial Ablation Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endometrial Ablation (4th gen) (Experimental): A single-centre uncontrolled observational study is proposed. All women presenting to the gynaecology outpatient clinic with heavy menstrual bleeding (HMB) in the absence of recognizable pelvic pathology, as determined by one or all of a normal pelvic ultrasound, hysteroscopy and / or endometrial biopsy, refractory to medical therapy that persists despite treatment with recommended pharmacological agents, who have no desire to preserve their fertility and are willing to have an endometrial ablation will be invited to participate. Eligible women with HMB will undergo RFA G4 endometrial ablation in either an inpatient or outpatient setting according to their preference.
  Interventions: Device: Endometrial ablation (4th gen)

INTERVENTIONS:
Device: Endometrial ablation (4th gen) — Radiofrequency Bipolar endometrial ablation device that is inserted into the uterine cavity to destroy the endometrial lining

SUMMARY:
All women presenting to the gynaecology outpatient clinic with heavy menstrual bleeding (HMB) in the absence of recognizable pelvic pathology, as determined by one or all of a normal pelvic ultrasound, hysteroscopy and / or endometrial biopsy, refractory to medical therapy that persists despite treatment with recommended pharmacological agents(1,2), who have no desire to preserve their fertility and are willing to have an endometrial ablation will be invited to participate. Eligible women with HMB will undergo radiofrequency G4 endometrial ablation in either an inpatient or outpatient setting according to their preference.

Outcomes will be assessed by administering postal questionnaires to measure menstrual bleeding symptoms including rates of amenorrhoea, dysmenorrhoea and life quality at baseline and at 6, and 12 months after ablative treatment. After the main study, there will be an additional evaluation of the long-term effects of outpatient ablative treatments of the endometrium by postal survey at 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Women with no desire to preserve their fertility who have heavy menstrual bleeding without organic pathology (DUB) of more than six months duration
2. Associated functional disability (negative impact on life quality).
3. Lack of response to medical treatment.
4. Prepared to undergo surgical treatment without general anaesthesia

Exclusion Criteria:

1. Women under 25 years
2. Suspected genital tract infection
3. Uterine pathology including endometrial pathology on endometrial biopsy (e.g. endometrial hyperplasia or carcinoma) and structural lesions (e.g. uterine malformations, adhesions, polyps, submucous fibroids or extracavity fibroids > 3cm in diameter) as identified on pelvic ultrasound and/or outpatient hysteroscopy.
4. Uterine cavity length >11cm
5. Adnexal pathology
6. Previous open myomectomy or endometrial ablation / resection and classical caesarian section
7. Patients considered vulnerable (e.g. current mental illness, emotionally labile, learning difficulties, immaturity)

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-03; Primary Completion 2015-10 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Amenorrhoea | 6 months
  Two Likert-type ordinal scales will be used to assess the change in menstrual blood loss using the questions and following response categories: 'How would you describe your menstrual periods?': 'No bleeding', 'Spotting or discharge only', 'Light bleeding', 'Moderate bleeding', 'Heavy bleeding' and 'Compared to before treatment, would you say that your heavy menstrual bleeding is: 'Much better, 'A little better', 'Same', 'Worse'. These scales will be administered in our study at 6, 12 and 60 months after the intervention.

SECONDARY OUTCOMES:
Visual analogue scale for assessment of pain | 6 months
  This technique involves use of 10 cm line on a piece of paper representing a continuum of the patients' opinion of the degree of pain. It is explained to the patient that the one extreme of the line represents "no pain at all" while the other represents "as much pain as she can possibly imagine". The subject rates the degree of pain by placing a mark on the line and scale values are obtained by measuring the distance from zero to that mark. The reliability of visual analogue scales in the assessment of pain has been established as reproducible and accurate. These scales will be administered in our study immediately following treatment, at one hour post treatment and on discharge from hospital.
Disease specific health-related quality of life | 6 months
  The multi-attribute utility assessment for menorrhagia questionnaire attempts to capture the consequences of menorrhagia on these domains with 6 questions each with 4 levels of response giving an overall composite score out of 100.

CONTACTS AND LOCATIONS:
Overall Officials: Justin Clark, MD, Principal Investigator — Birmingham Women's NHS Foundation Trust

REFERENCES:
- [Background] 1. Royal College of Obstetricians and Gynaecologists. The initial management of menorrhagia. Evidence-Based Clinical Guideline No.4.London: RCOG Press; 1999.
- [Background] 2. Royal College of Obstetricians and Gynaecologists. The Management of Menorrhagia in Secondary Care. Evidence-Based Clinical Guideline No.5.London: RCOG Press; 1999.